CLINICAL TRIAL: NCT06166758
Title: Pilot Feasibility Study: Educational Genetic Test Video
Brief Title: Feasibility Study: Educational Genetic Test Video
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MCC-23-20539; HM20028425 (Other: Virginia Commonwealth University)
Record Dates: First submitted 2023-12-01; First posted 2023-12-12 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Prostate Cancer; Education
Keywords: Genetic testing education
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Educational Video (Experimental): Educational video about germline genetic testing, which is 7 minutes long
  Interventions: Behavioral: Educational Video

INTERVENTIONS:
Behavioral: Educational Video — Educational video regarding the benefits, risks, and limitations of genetic testing for hereditary cancer risk.

SUMMARY:
Assess whether introducing an educational video regarding the benefits, risks, and limitations of genetic testing affects prostate cancer patients' decisional conflict regarding receiving germline genetic testing.

ELIGIBILITY:
Inclusion Criteria:

* Prostate cancer patients who have been prescribed germline genetic testing by their provider
* Understand written and spoken English
* Have not received germline genetic testing for hereditary cancer risk in the past

Exclusion Criteria:

* Adults unable to consent
* Individuals who are not yet adults (infants, children, teenagers)
* Pregnant individuals
* Prisoners

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2023-12-14 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
Assess the value of presenting patients an educational video regarding the benefits risks, and limitations of genetic testing for hereditary cancer risk. | Day 1
  Determine proof-of concept by the results of a patient survey to assess the effect that the video has on decisional conflict. The survey administered post intervention uses a modified decisional conflict scale in a pre then post format. This is a 5 point Likert scale where 1 equals no, 2= probably no, 3= unsure, 4= probably yes, and 5=yes. This format asks participants to imagine their thoughts on the subject before having watched the video, then to clarify their thoughts on the same subjects now that they have watched the video.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Monast, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
There are no plans to share individual participant data.